CLINICAL TRIAL: NCT06441201
Title: Peripheral Pulse Volume Changes in Acute Gastrointestinal Bleeding
Brief Title: Acute Gastrointestinal Bleeding Peripheral Pulse Volume Changes
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jad P. AbiMansour, Principal Investigator, Mayo Clinic
Other Study IDs: 23-005579
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: GastroIntestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastrointestinal Bleeding Peripheral Pulse Volume: Subject undergoing an emergency endoscopic evaluation for active gastrointestinal bleeding will have their peripheral pulse volumes monitored using a pulse flowmeter throughout the procedure and 2 hours after the procedure.
  Interventions: Diagnostic Test: Pulse flowmeter

INTERVENTIONS:
Diagnostic Test: Pulse flowmeter — Measures peripheral pulse volumes by an electrode applied non-invasively to the lower extremity (left or right) at the beginning of the endoscopic evaluation for the duration of the procedure, and up to 2 hours after the completion of the procedure.

SUMMARY:
The purpose and aim of this study are to compare changes in pulse volume to non-invasively predict active bleeding or high-risk stigmata in patients undergoing a gastrointestinal endoscopy to assess feasibility of the flow meter clinically.

DETAILED DESCRIPTION:
The maximum change in volume of a limb segment during the cardiac cycle - pulse volume - will be monitored non-invasively along with standard vitals in patients with a suspected gastrointestinal bleed undergoing endoscopy. Pulse volume and vitals will be collected prior to and following endoscopy up to the point of dismissal from the endoscopy unit so that the data may be correlated with the endoscopic and clinical findings.

ELIGIBILITY:
Inclusion Criteria:

- Adults (age >18yr) undergoing emergent endoscopy for active GI bleeding.

Exclusion Criteria:

* Patients with pre-existing heart failure (ejection fraction <40%), cardiac rhythm abnormalities and peripheral vascular disease.
* Patients with underlying implanted cardiac electrical devices and spinal cord stimulators.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing emergent endoscopic evaluation for active gastrointestinal bleeding at Mayo Clinic, Rochester, Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Changes in peripheral pulse volume with and without active bleeding | Baseline, approximately 2 hours post endoscopy
  Peripheral pulse volume as measured by pulse flowmeter (uL/cm) pre and post endoscopic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Storm, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No